CLINICAL TRIAL: NCT02721628
Title: Femtosecond Laser Assisted Epi-keratoplasty Versus Collagen Cross-Linking in Progressive Keratoconus
Brief Title: Epi-keratoplasty Versus Collagen Cross-Linking in Progressive Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gao Xinbo, Attendant Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zoc-ekccl2015
Record Dates: First submitted 2016-03-06; First posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Progressive Keratoconus
Keywords: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epi-keratoplasty Group (Experimental): Epi-keratoplasty Group: Reversible keratoplasty performed with only the removal of corneal epithelium of the host cornea. A donor graft is transplanted on the recipients' eye locating on the Bowman's layer.
  Interventions: Procedure: Epi-keratoplasty; Device: Femtosecond laser
- Collagen Cross-Linking Group (Active Comparator): Collagen Cross-Linking: Corneal epithelium is mechanically removed. Then, a solution of riboflavin is instilled each minute for 30 minutes. Corneas are irradiated by a UVA light for 3mW/cm2 during 30 minutes
  Interventions: Procedure: Collagen Cross-Linking

INTERVENTIONS:
Procedure: Epi-keratoplasty — Femtosecond laser assisted Epi-keratoplasty
  Arms: Epi-keratoplasty Group
Procedure: Collagen Cross-Linking — Collagen Cross-Linking: Standard procedure, which is descriptor bellows: Corneal epithelium is mechanically removed. Then, a solution of riboflavin is instilled each minute for 30 minutes. Corneas are irradiated by a UVA light for 3mW/cm2 during 30 minutes
  Other Names: CCL
  Arms: Collagen Cross-Linking Group
Device: Femtosecond laser — Use in the epic-keratoplasty surgery
  Arms: Epi-keratoplasty Group

SUMMARY:
Epi-keratoplasty Versus Collagen Cross-Linking in Progressive Keratoconus

DETAILED DESCRIPTION:
Keratoconus is a bilateral corneal ecstatic disease which is not uncommon and always behaves progressively and results in visual impairment by inducing irregular astigmatism and corneal opacities.

Collagen Cross-Linking (CXL) is widely used in progressive keratoconus. The cornea is soaked with a riboflavin solution and then being exposed to ultraviolet-A radiation. The performance creates links between collagen fibrils in order to rigidify the corneal stroma and slow down the progression of keratoconus. However, the effectiveness is not satisfied and accompanied with risks of side effects and serious complications, such as pain for the first two post-operative days, temporary loss of visual acuity during the first three months, infection and stromal opacity due to corneal scarring.

Epi-keratoplasty is a reversible technique in which a corneal graft is transplanted on the recipients' eye with only removal of the epithelium of the receptor cornea. The procedure was assisted by femtosecond laser which allows precisely and neatly cutting. The graft strengths the whole host corneal rigidity and roughness and therefore renders the progression of keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Keratoconus
* Age ≥ 18 years old
* Corneal thickness ≥ 400 µm
* Progressive stage 1 to 3 keratoconus (Krumeich classification)

Exclusion Criteria:

* Corneal thickness < 400µm
* Concomitant corneal disease
* History of corneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Changes of Spherical equivalent | 01012016~01012018: preoperatively, postoperatively 2 weeks, 1,2,3,6,12 months, 2 years

SECONDARY OUTCOMES:
maximum keratometry (K-max) derived from computerized video keratography | 01012016~01012018: preoperatively, postoperatively 2 weeks, 1,2,3,6,12 months, 2 years
minimum keratometry | 01012016~01012018: preoperatively, postoperatively 2 weeks, 1,2,3,6,12 months, 2 years
  also from computerized video keratography, the opposite description of K-max
Visual acuity | 01012016~01012018: preoperatively, postoperatively 2 weeks, 1,2,3,6,12 months, 2 years

OTHER OUTCOMES:
Spherical equivalent | 01012016~01012018: preoperatively, postoperatively 2 weeks, 1,2,3,6,12 months, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- ZhongShan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided